CLINICAL TRIAL: NCT02151188
Title: Liquid Protein Preloads With Different Carbohydrate Types Effects on the Glycaemic and Insulinaemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Associate Professor, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014/00036
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes; Impaired Glucose Tolerance; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Obesity | interventions — Bread; Soy Milk; Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Bread and water (Other): co-ingestion control session
  Interventions: Dietary Supplement: Bread, Soy milk and cow milk; Device: real-time ultrasonography (GE LOGIQ P5 ultrasound in CNRC)
- bread with cow milk co-ingestion (Experimental): co-ingestion bread with cow milk
  Interventions: Dietary Supplement: Bread, Soy milk and cow milk; Device: real-time ultrasonography (GE LOGIQ P5 ultrasound in CNRC)
- bread with soy milk co-ingestion (Experimental): co-ingestion bread with soy milk
  Interventions: Dietary Supplement: Bread, Soy milk and cow milk; Device: real-time ultrasonography (GE LOGIQ P5 ultrasound in CNRC)
- preload cow milk (Experimental): preload cow milk 30 min, then bread
  Interventions: Dietary Supplement: Bread, Soy milk and cow milk; Device: real-time ultrasonography (GE LOGIQ P5 ultrasound in CNRC)
- preload soy milk (Experimental): preload soy milk 30 min, then bread
  Interventions: Dietary Supplement: Bread, Soy milk and cow milk; Device: real-time ultrasonography (GE LOGIQ P5 ultrasound in CNRC)

INTERVENTIONS:
Dietary Supplement: Bread, Soy milk and cow milk — The study will examine the metabolic effects of two liquid proteins (soy milk and cow milk) with carbohydrate (bread) meals.
Device: real-time ultrasonography (GE LOGIQ P5 ultrasound in CNRC)

SUMMARY:
This study hypothesizes that milk protein consumed together or shortly before a white rice or white bread carbohydrate meal exerts different influence on the glycaemic, insulinaemic responses.

DETAILED DESCRIPTION:
Consumption of milk proteins increase satiety and reduce glucose response when consumed alone or with carbohydrate. Milk proteins are of interest because proteins are more satiating than either carbohydrate or fat, and they regulate food intake and metabolic functions by the intact protein, encrypted peptides and amino acids on gastrointestinal and central pathways. White rice and white bread are two common carbohydrates types mostly consumed in Asia. Both of them are known to result in high glycaemic and insulinaemic responses. However, in most meals, they are accompanied by other foods such as soy milk, cow milk products. The glyceamic and insulinaemic responses are determined by the type of protein and the type of carbohydrates. And also the consumption time of protein and carbohydrate. Recent research points to an intrinsic value of small amounts of milk protein or dairy consumed shortly before a meal can reduce the glycemic response to carbohydrate and that this is not at the cost of increased demand for insulin. The objective of the present study is to investigate how glycaemic, insulinaemic and satiety responses to a white rice or white bread meal changed when a soy milk or cow milk consumed together or shortly before the meal. Whole soy milk and whole cow milk will be added to the meal. Healthy subjects (n 15) will ingest the test meals once. The meals will be provided as breakfasts, on 10 different occasions, in random order with ≥ 7 days between each. Blood samples (from the cannula and finger pricks) will be then drawn for 3 h, and glucose and serum insulin, plasma glucagon, satiety markers, inflammation markers, amino acids et.al will be analysed. The objective of the study is determining if different liquid protein consumed shortly before or with carbohydrate has different effects on metabolism. And also we will compare the difference of white rice and white bread. Determining the consuming time effect, milk protein type and carbohydrate type on glycaemic and insulinaemic are critical for the provision of dietary advice and formulation of public health guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Age between 21-40 years
* Not on prescription medication known to affect glucose and satiety related metabolism
* Do not partake in sports at the competitive and/or endurance levels
* Weight of at least 45kg
* Body mass index between 18.0 to 24.9 kg/m2
* Normal blood pressure (120/80 mmHg)

Exclusion Criteria: Smoker

* fasting blood glucose>5.5 mmol/L
* Any major medical conditions including diabetes, hypertension, cardiovascular disease, thyroid disorders
* Allergic or intolerant to foods presented in the study

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glucose response of different treatments | 3.5 hrs post consumption
  The blood glucose will be measured by Hemocue 201 from finger prick. Venous blood will be collected at the same time points.

SECONDARY OUTCOMES:
Gastric emptying rate | 2 hours post consumption
  Measurement of gastric emptying rate using real-time ultrasonography (GE LOGIQ P5 ultrasound in CNRC). Ultrasound measurements will be taken with subjects in a supine position during fasting, then at 15-30 min intervals after consumption of the test meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

REFERENCES:
- [Derived] Sun L, Tan KWJ, Han CMS, Leow MK, Henry CJ. Impact of preloading either dairy or soy milk on postprandial glycemia, insulinemia and gastric emptying in healthy adults. Eur J Nutr. 2017 Feb;56(1):77-87. doi: 10.1007/s00394-015-1059-y. Epub 2015 Oct 6. PMID 26439722